CLINICAL TRIAL: NCT01337869
Title: Comparison of Bascom Cleft Lift Technique Versus Limberg Flap Closure for Treatment of Sacrococcygeal Pilonidal Disease: A Prospective Randomized Controlled Trial Evaluating for Patient Satisfaction and Early Recurrence
Brief Title: Bascom Cleft Lift Versus Limberg Flap for Sacrococcygeal Pilonidal Sinus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trabzon Numune Training and Research Hospital (Other Government)
Responsible Party: Ali GUNER, M.D., Trabzon Numune Training and Research Hospital, Department of General Surgery
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TNEAH-2010GC1
Record Dates: First submitted 2011-04-15; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Pilonidal Sinus
Keywords: Bascom Procedure, Limberg, Pilonidal Disease
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bascom Cleft Lift Technique (Active Comparator)
  Interventions: Procedure: Bascom Cleft Lift
- Limberg Flap Technique (Active Comparator)
  Interventions: Procedure: Limberg Flap

INTERVENTIONS:
Procedure: Bascom Cleft Lift — Patients are positioned prone. The skin incision is drawn on the natal cleft, marking out the area of skin to be excised. The skin from this side of the natal cleft is then elevated. The skin on the opposite side of the cleft then is undermined to a distance required to allow primary closure of the defect away from the midline without tension. The elevated skin island is excised. The sinuses remaining in the deeper tissues are curetted thoroughly. Hemostasis is maintained. A 12F low-suction drain is sited and fat of the natal cleft then is approximated by using an absorbable suture. The wound is closed with a 3-0 polypropylene suture.The drain remains in situ to time that drainage amount decreases below 20 ml/day. The suture is removed in the clinic 10 day after surgery.
  Other Names: Bascom Procedure
  Arms: Bascom Cleft Lift Technique
Procedure: Limberg Flap — Patients are positioned prone. The area to be excised is mapped-out, and the flap is designed. The area to be excised is mapped on the skin in a rhomboid form. The skin incision is deepened to the presacral fascia. Tissue is removed en bloc. After removing the rhombic excision, the Limberg fascia cutaneous flap is prepared through the right or left-side gluteus maximus fascia. The flap is fully mobilized and transposed medially to fulfill the rhombic defect without any tension. Hemosthasis is accomplished. A 12F low-suction drain is sited and wound is closed in two layers: the subcutaneous tissue with absorbable suture and the skin with 3/0 polypropylene. drain remains in situ to time that drainage amount decreases below 20 ml/day. The suture is removed in the clinic 10 day after surgery.
  Other Names: Limbergplasty
  Arms: Limberg Flap Technique

SUMMARY:
A pilonidal sinus is a cyst on the natal cleft of the buttocks that often contains hair and skin debris. The condition is common and requires surgery to be cured. Several surgical procedures are described in literature. Limberg Flap technique is frequently used technique for this disease all over the world. However, Bascom Cleft Lift Technique is relatively newer technique. The purpose of this prospective randomized study is comparison of these techniques about patient satisfaction for postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* All types of pilonidal sinus or cyst
* The patient understands trial information and is capable of making a decision for informed consent after having received information.
* The patient wants to undergo surgery for pilonidal sinus and accepts participation in the trial.

Exclusion Criteria:

* acute abscess formation (Cruse-Foord Class IV)
* patient with minor inflammation are included to trial after two-week antibiotic treatment (Cruse-Foord Class III)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life and postoperative pain | within 30 days
  Determine patient satisfaction factors using the quality of life survey (SF-36 form) on the 10th-30th day and postoperative pain by using post-operative visual analog pain scale on the 2nd-10th day

SECONDARY OUTCOMES:
early recurrence rate | up to 6 months
  participants will be followed for the duration of hospital stay and first 30 days, up to 6 months. at the end of the study, recurrence rates will be presented for both groups.
Healing time | within 30 days
  determine wound healing time. the time until complete recovery will be presented.
operative time | during surgical procedure (day 1)
  the time between the beginning of the procedure and last skin suture.
hospital stay | during first week (one week)
  the time to until discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Trabzon Numune Training and Research Hospital, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Background] Bascom J, Bascom T. Failed pilonidal surgery: new paradigm and new operation leading to cures. Arch Surg. 2002 Oct;137(10):1146-50; discussion 1151. doi: 10.1001/archsurg.137.10.1146. PMID 12361421
- [Background] Mentes O, Bagci M, Bilgin T, Ozgul O, Ozdemir M. Limberg flap procedure for pilonidal sinus disease: results of 353 patients. Langenbecks Arch Surg. 2008 Mar;393(2):185-9. doi: 10.1007/s00423-007-0227-9. Epub 2007 Sep 22. PMID 17899165
- [Background] Nordon IM, Senapati A, Cripps NP. A prospective randomized controlled trial of simple Bascom's technique versus Bascom's cleft closure for the treatment of chronic pilonidal disease. Am J Surg. 2009 Feb;197(2):189-92. doi: 10.1016/j.amjsurg.2008.01.020. Epub 2008 Jul 17. PMID 18639221
- [Background] Jamal A, Shamim M, Hashmi F, Qureshi MI. Open excision with secondary healing versus rhomboid excision with Limberg transposition flap in the management of sacrococcygeal pilonidal disease. J Pak Med Assoc. 2009 Mar;59(3):157-60. PMID 19288942